CLINICAL TRIAL: NCT05079100
Title: Effectiveness of Counseling on Attitude and Use of Postpartum Family Planning Within 6 Weeks.
Brief Title: Effectiveness of Counseling on Use of Postpartum Family Planning.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Ismail Mohamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ECAUPFP
Record Dates: First submitted 2021-09-14; First posted 2021-10-15 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of intervention (counseling) (Active Comparator): the group will receive the contraception counseling
  Interventions: Other: postpartum contraception method counselling
- group of control (no counseling) (No Intervention): this group will not receive any counseling

INTERVENTIONS:
Other: postpartum contraception method counselling — It will be face-to-face counseling with females about the use of postpartum contraception methods within 6 weeks postpartum.
  Arms: group of intervention (counseling)

SUMMARY:
Family planning (FP) is the most supported, reasonable public health service to prevent both maternal and newborn mortality and decrease the risk of adverse maternal, perinatal, and infant outcomes. The World Health Organization's (WHO) recommend of waiting at least 2 years after a live birth before attempting the next pregnancy as short interval between pregnancies increase risk of preterm labor; low birth weight; fetal, early neonatal and infant death; and serious maternal outcomes.

DETAILED DESCRIPTION:
So WHO recommends postpartum family planning (PPFP) for healthy birth spacing. PPFP is divided into three stages immediate: within 48 hours following delivery, early: within the first 6 weeks after delivery, late: within 12 months postpartum. Fertility can return as soon as 45 days after delivery for non-breastfeeding women, and among women who are not breastfeeding exclusively, fertility can return before the return of menses. Providing PPFP instantaneously following delivery may be likeable for women who prefer effective postpartum protection as the return of fertility may be hard to expect. So Promoting PPFP use was documented in different communities, interventions included conversational, SMS, brochure and video-based contraceptive education in antenatal or postnatal visits. However, the unmet need for FP is high in the postpartum period, ranging from 32 to 62% in low and middle-income countries depending on the definition used. that is why WHO recommends that all women should be offered counselling within 6 weeks postpartum so we will study the impact of post-partum counselling pre and post-discharge on intent and use of a reliable family planning method.

ELIGIBILITY:
Inclusion Criteria:

1. Women who delivered in Women's Health hospitals, Assiut university hospitals.
2. Women in reproductive age (15 - 49 years).
3. Accepting to share in our study.

Exclusion Criteria:

1. Women diagnosed with mental problems or postpartum psychosis
2. Women with unstable hemodynamic status.
3. Women after Peripartum hysterectomy or tubal ligation.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
number of participant will Use postpartum contraception methods | 6 weeks
  we will study by questionnaire in interview session the number of participants who will use postpartum contraception methods within 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Galal Mahran, Prof, Study Director — Department of public health and community medicine, Faculty of medicine, Assiut university.
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gul X, Hameed W, Hussain S, Sheikh I, Siddiqui JU. A study protocol for an mHealth, multi-centre randomized control trial to promote use of postpartum contraception amongst rural women in Punjab, Pakistan. BMC Pregnancy Childbirth. 2019 Aug 8;19(1):283. doi: 10.1186/s12884-019-2427-z. PMID 31395034
- [Background] Cooper CM, Charurat E, El-Adawi I, Kim YM, Emerson MR, Zaki W, Schuster A. Postpartum Family Planning During Sociopolitical Transition: Findings from an Integrated Community-Based Program in Egypt. Int Perspect Sex Reprod Health. 2016 Jun 1;42(2):57-69. doi: 10.1363/42e1216. PMID 28825907
- [Background] Pradhan E, Canning D, Shah IH, Puri M, Pearson E, Thapa K, Bajracharya L, Maharjan M, Maharjan DC, Bajracharya L, Shakya G, Chaudhary P. Integrating postpartum contraceptive counseling and IUD insertion services into maternity care in Nepal: results from stepped-wedge randomized controlled trial. Reprod Health. 2019 May 29;16(1):69. doi: 10.1186/s12978-019-0738-1. PMID 31142344
- [Background] Burapasikarin C, Manonai J, Wattanayingcharoenchai R. The effect of an educational video on long-acting reversible contraception (LARC) utilization at 6-8 weeks postpartum period: a randomized controlled trial. Arch Gynecol Obstet. 2020 Dec;302(6):1503-1509. doi: 10.1007/s00404-020-05710-3. Epub 2020 Jul 30. PMID 32734413
- [Background] Tang JH, Dominik RC, Zerden ML, Verbiest SB, Brody SC, Stuart GS. Effect of an educational script on postpartum contraceptive use: a randomized controlled trial. Contraception. 2014 Aug;90(2):162-7. doi: 10.1016/j.contraception.2014.03.017. Epub 2014 Apr 12. PMID 24833047
- [Background] Harrington EK, Drake AL, Matemo D, Ronen K, Osoti AO, John-Stewart G, Kinuthia J, Unger JA. An mHealth SMS intervention on Postpartum Contraceptive Use Among Women and Couples in Kenya: A Randomized Controlled Trial. Am J Public Health. 2019 Jun;109(6):934-941. doi: 10.2105/AJPH.2019.305051. PMID 31067089